CLINICAL TRIAL: NCT04145440
Title: A Phase Ib/IIa, Open-Label, Multicenter Clinical Trial to Assess Safety and Efficacy of the Human Anti-CD38 Antibody MOR202 in Anti-PLA2R Antibody Positive Membranous Nephropathy (aMN)
Brief Title: Trial to Assess Safety and Efficacy of MOR202 in Anti-PLA2R + Membranous Nephropathy (aMN)
Acronym: M-PLACE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HI-Bio, A Biogen Company (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR202C103
Record Dates: First submitted 2019-10-18; First posted 2019-10-30 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Glomerulonephritis, Membranous; antiPLA2R Positive
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — felzartamab

STUDY DESIGN:
Intervention Model Description: 2 cohorts by disease status (Cohort 1: Patients with newly diagnosed or relapsed membranous nephropathy; Cohort 2: Patients with membranous nephropathy refractory to immunosuppressive treatment)
Masking Description: The study is open label as all patients receive the same Investigational Medicinal Product (IMP) and same dose
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (newly diagnosed or relapsed participants) (Experimental): Participants with newly diagnosed or relapsed membranous nephropathy received MOR202 as an intravenous infusion over 6 treatment cycles of 28-days each. Dosing occurred weekly in Cycle 1 and every 4 weeks in Cycles 2 to 6.
  Interventions: Drug: MOR202
- Cohort 2 (refractory participants) (Experimental): Participants with membranous nephropathy refractory to immunosuppressive treatment received MOR202 as an intravenous infusion over 6 treatment cycles of 28-days each. Dosing occurred weekly in Cycle 1 and every 4 weeks in Cycles 2 to 6.
  Interventions: Drug: MOR202

INTERVENTIONS:
Drug: MOR202 — Patients received 9 doses of MOR202 as an intravenous infusion over 6 treatment cycles of 28-days each. Dosing occured weekly in Cycle 1 and every 4 weeks in Cycles 2 to 6.

SUMMARY:
This is an open-label, multicentre study to characterize the safety and efficacy of the human anti-CD38 antibody MOR202 in adult subjects with in Anti-PLA2R Antibody Positive Membranous Nephropathy (newly diagnosed/relapsed/refractory)

DETAILED DESCRIPTION:
After treatment subjects will be observed for up to 1 year.

Study Sponsor, originally HI-Bio, Inc., is now HI-Bio, A Biogen Company.

ELIGIBILITY:
Key Inclusion Criteria:

* > 18 to < 80 years (at date of signing informed consent form [ICF]).
* Urine protein to creatinine ratio (UPCR) of ≥ 3.000 g/g OR proteinuria ≥ 3.500 g/24 h from 24-h urine at screening
* Active anti-PLA2R antibody positive MN in need of immunosuppressive therapy (IST) according to investigator judgement and diagnosed on the basis of a biopsy, archival biopsy acquired within 5 years prior to screening is acceptable.
* Estimated glomerular filtration rate ≥ 50 ml/min/1.73m² or ≥ 30 and <50 ml/min/1.73m², and interstitial fibrosis and tubular atrophy score of less than 25% on a renal biopsy obtained within the last 6 months prior to start of screening.
* Not in spontaneous remission despite proper treatment with ACEIs, ARBs (sufficient dose and treatment duration) as per clinical practice and scientific guidelines. If the subject is intolerant to an ACEI or ARB, the reason must be documented and approval obtained prior to enrolment.
* Systolic blood pressure BP ≤150 mmHg and diastolic BP ≤100 mmHg after 5 minutes of rest
* Vaccinated against Pneumococcus within the last 5 years prior to date of signing informed consent (subjects may be vaccinated during screening to meet this criterion; interval to first dose of MOR202 must be at least 14 days).
* Cohort 1 comprises newly diagnosed or relapsed subjects: Serum anti-PLA2R antibodies ≥50.0 RU/mL
* Cohort 2 comprises therapy refractory subjects: a Subject did not achieve immunological remission after prior IST(s) as documented by the investigator AND b Subject is without promising standard therapeutic options as documented by the investigator (i.e. investigator expects efficacy or safety issues with remaining IST options) AND c Serum anti-PLA2R antibodies ≥ 20.0 RU/mL measured at screening

Note: France will only enroll patients in Cohort 2.

Key Exclusion Criteria:

* Hemoglobin < 80 g/L.
* Thrombocytopenia: Platelets < 100.0 x 109/L.
* Neutropenia: Neutrophils < 1.5 x 109/L.
* Leukopenia: Leukocytes < 3.0 x 109/L.
* Hypogammaglobulinemia: Serum immunoglobulins ≤ 4.0 g/L.

Subjects may receive supportive therapies to meet the above criteria

* B-cells < 5 x 106/L.
* Secondary cause of MN (e.g. Systemic lupus erythematosus, medications, malignancies)
* Concomitant renal disease other than MN (e.g., diabetic renal disease, lupus nephritis, IgA nephropathy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — HI-Bio, A Biogen Company
Locations (45):
- United States (11):
  - North America Research Institute, Azusa, California
  - UCSF Medical Center, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - University of Miami Division of Nephrology & Hypertension, Miami, Florida
  - GA Nephrology Associates, Lawrenceville, Georgia
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - Kidney Care and Transplant Services of New England, PC, Springfield, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - MedResearch, Inc, El Paso, Texas
  - Texas Research Institute, Fort Worth, Texas
- Australia (3):
  - St. George Hospital, Sydney, New South Wales
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western Health, Melbourne
- Belgium (6):
  - O.L.V. Ziekenhuis, Aalst
  - C.H.U. Brugmann - Site Victor Horta, Brussels
  - Universitair Ziekenhuis Brussels, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- France (5):
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - Hopital Claude Huriez -CHU Lille, Lille
  - Hopital Tenon Service de nephrologie, Paris
  - CHU Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Ospedale Borgo Roma, Verona
- Radboud UMC Niimegen Nephrology, Nijmegen, Netherlands
- Poland (3):
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Centrum Zdrowia MDM, Warsaw
  - Miedzyleski Szpital Specjalistyczny, Warsaw
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 65 participants were screened for this study. 31 participants were enrolled and received at least one dose of study drug.
Period: Overall Study
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Started | 18 | 13
Received at Least 1 Dose of Study Drug | 18 | 13
Completed | 13 | 10
Not Completed | 5 | 3
Not completed — Physician Decision | 3 | 0
Not completed — Use of prohibited therapy | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants) | Total
Number analyzed (Participants) | 18 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.34) | 55.0 (12.47) | 57.5 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 16 | 8 | 24
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 1 to Week 24
Population: The Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
Participants | 15 | 12

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 1 to Week 24
Population: The Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
percentage of participants | 83.3 | 92.3

3. Secondary Outcome: Best Immunological Response Rate (BIRR)
Description: The BIRR was defined as the percentage of participants with a best immunological response of stringent immunological complete response (sICR), immunological complete response (ICR), or immunological partial response (IPR) prior to the start of prohibited treatment or progression, based on reduction of serum anti-PLA2R antibody titer.
Time Frame: Up to 52 weeks
Population: The FAS included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
percentage of participants | 83.3 [58.6 to 96.4] | 61.5 [31.6 to 86.1]

4. Secondary Outcome: Number of Participants Tested Positive for Anti-felzartamab Antibodies
Time Frame: Baseline; Up to 52 weeks
Population: The Immunogenicity Analysis Set (IAS) included all participants with at least one antidrug antibody (ADA) result available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 15 | 13
Participants
  Baseline | 1 | 1
  Post First Dose (52 weeks) | 1 | 0

5. Secondary Outcome: Percentage of Participants Tested Positive for Anti-felzartamab Antibodies
Time Frame: Baseline; Up to 52 weeks
Population: The IAS included all participants with at least one ADA result available.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 15 | 13
percentage of participants
  Baseline | 6.7 | 7.7
  Post First Dose (52 weeks) | 6.7 | 0.0

6. Secondary Outcome: Antibody Titers of Participants Tested Positive for Anti-felzartamab Antibodies
Time Frame: Baseline; Up to 52 weeks
Population: The IAS included all participants with at least one ADA result available. Here, the "Overall Number of Participants Analyzed" equals the number of participants with positive ADA titers and "Number Analyzed" is the number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: anti-felzartamab antibody titers
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 1 | 1
anti-felzartamab antibody titers
  Baseline | 13.10 (NA) — Standard deviation not calculable with n=1 | 11.50 (NA) — Standard deviation not calculable with n=1
  Post First Dose (52 weeks): number analyzed (Participants) | 1 | 0
  Post First Dose (52 weeks) | 3.48 (NA) — Standard deviation not calculable with n=1 |

7. Secondary Outcome: Felzartamab Serum Concentrations After Multiple Intravenous Administrations
Time Frame: Pre Dose and Post Dose on Cycle 1 Day 1 (C1D1), C1D8, C1D15, C1D22, C2D1, C3D1, C4D1, C5D1, C6D1, End of Treatment (week 24), Follow-up visit (week 38), End of Study (up to 52 weeks)
Population: The Pharmacokinetic Analysis Set (PKAS) included all participants with evaluable felzartamab serum concentration data. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and the "Number Analyzed" shows the number of participants evaluated at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram(s)/millilitre (ng/mL)
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
nanogram(s)/millilitre (ng/mL)
  Pre-dose C1D1 | 0.0 (0.0) | 0.0 (0.0)
  Post-dose C1D1 | 323499.3 (98.3) | 301417.5 (151.9)
  Pre-dose C1D8: number analyzed (Participants) | 17 | 11
  Pre-dose C1D8 | 89381.7 (97.9) | 129924.9 (100.7)
  Post-dose C1D8: number analyzed (Participants) | 17 | 11
  Post-dose C1D8 | 425669.4 (50.7) | 429629.4 (91.7)
  Pre-dose C1D15: number analyzed (Participants) | 17 | 12
  Pre-dose C1D15 | 174658.7 (75.5) | 189047.7 (80.9)
  Post-dose C1D15: number analyzed (Participants) | 16 | 12
  Post-dose C1D15 | 456390.9 (70.6) | 547940.5 (60.2)
  Pre-dose C1D22: number analyzed (Participants) | 17 | 11
  Pre-dose C1D22 | 185140.7 (78.0) | 286607.9 (25.7)
  Post-dose C1D22: number analyzed (Participants) | 17 | 10
  Post-dose C1D22 | 495612.5 (57.3) | 656862.8 (29.7)
  Pre-dose C2D1: number analyzed (Participants) | 17 | 12
  Pre-dose C2D1 | 24903.4 (47.3) | 148097.2 (193.7)
  Post-dose C2D1: number analyzed (Participants) | 16 | 11
  Post-dose C2D1 | 474157.9 (108.0) | 415814.9 (106.3)
  Pre-dose C3D1: number analyzed (Participants) | 17 | 12
  Pre-dose C3D1 | 34111.0 (164.7) | 25879.8 (572.2)
  Pre-dose C4D1: number analyzed (Participants) | 13 | 11
  Pre-dose C4D1 | 19811.2 (218.1) | 30655.9 (128.9)
  Pre-dose C5D1: number analyzed (Participants) | 14 | 9
  Pre-dose C5D1 | 27021.6 (152.0) | 35176.1 (84.1)
  Pre-dose C6D1: number analyzed (Participants) | 14 | 8
  Pre-dose C6D1 | 28734.6 (116.9) | 30383.0 (88.8)
  End of Treatment (week 24): number analyzed (Participants) | 17 | 10
  End of Treatment (week 24) | 12367.0 (349.9) | 33813.6 (61.9)
  Follow-up visit (week 38): number analyzed (Participants) | 1 | 0
  Follow-up visit (week 38) | 369.0 (NA) — Geometric %CV not calculable with n=1 |
  End of Study (up to week 52): number analyzed (Participants) | 1 | 0
  End of Study (up to week 52) | 278.0 (NA) — Geometric %CV not calculable with n=1 |

8. Secondary Outcome: Number of Participants With AEs During the Follow-up Period
Description: as for outcome 2
Time Frame: Week 25 to Week 52
Population: The Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
Participants | 8 | 5

9. Secondary Outcome: Percentage of Participants With AEs During the Follow-up Period
Description: as for outcome 2
Time Frame: Week 25 to Week 52
Population: The Safety Analysis Set included all participants who received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) | Cohort 2 (Refractory Participants)
Number analyzed (Participants) | 18 | 13
percentage of participants | 44.4 | 38.5

ADVERSE EVENTS:
Time Frame: Week 1 to Week 52 (Weeks 1-24 [Treatment Period]; Weeks 25-52 [Follow-up Period])
Description: The Safety Analysis Set included all participants who received at least one dose of study drug. As pre-specified, data are presented split for the treatment period and follow-up period.
Groups:
- Cohort 1 (Newly Diagnosed or Relapsed Participants) Treatment Period (Weeks 1-24): Participants with newly diagnosed or relapsed membranous nephropathy received MOR202 as an intravenous infusion over 6 treatment cycles of 28-days each. Dosing occurred weekly in Cycle 1 and every 4 weeks in Cycles 2 to 6.
- Cohort 2 (Refractory Participants) Treatment Period (Weeks 1-24): Participants with membranous nephropathy refractory to immunosuppressive treatment received MOR202 as an intravenous infusion over 6 treatment cycles of 28-days each. Dosing occurred weekly in Cycle 1 and every 4 weeks in Cycles 2 to 6.
- Cohort 1 (Newly Diagnosed or Relapsed Participants) Follow-up Period (Weeks 25-52): Participants with newly diagnosed or relapsed membranous nephropathy.
- Cohort 2 (Refractory Participants) Follow-up Period (Weeks 25-52): Participants with membranous nephropathy refractory to immunosuppressive treatment.
Arm/Group | Cohort 1 (Newly Diagnosed or Relapsed Participants) Treatment Period (Weeks 1-24) | Cohort 2 (Refractory Participants) Treatment Period (Weeks 1-24) | Cohort 1 (Newly Diagnosed or Relapsed Participants) Follow-up Period (Weeks 25-52) | Cohort 2 (Refractory Participants) Follow-up Period (Weeks 25-52)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/13 | 0/18 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/13 | 1/18 | 1/13
Other Adverse Events (participants affected / at risk) | 15/18 | 12/13 | 8/18 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Newly Diagnosed or Relapsed Participants) Treatment Period (Weeks 1-24) (N=18) | Cohort 2 (Refractory Participants) Treatment Period (Weeks 1-24) (N=13) | Cohort 1 (Newly Diagnosed or Relapsed Participants) Follow-up Period (Weeks 25-52) (N=18) | Cohort 2 (Refractory Participants) Follow-up Period (Weeks 25-52) (N=13)
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Newly Diagnosed or Relapsed Participants) Treatment Period (Weeks 1-24) (N=18) | Cohort 2 (Refractory Participants) Treatment Period (Weeks 1-24) (N=13) | Cohort 1 (Newly Diagnosed or Relapsed Participants) Follow-up Period (Weeks 25-52) (N=18) | Cohort 2 (Refractory Participants) Follow-up Period (Weeks 25-52) (N=13)
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 0 | 1
Chest pain (General disorders) | 1 | 2 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Vaccination site pain (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 7 | 1 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 3 | 0 | 1 | 0
Lymphocyte percentage decreased (Investigations) | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Monocyte count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 8 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Decreased appetite (Nervous system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 4 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hypoferritinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04145440/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT04145440/SAP_001.pdf